CLINICAL TRIAL: NCT06632093
Title: Hepatic Arterial Infusion Chemotherapy in Combination with PD-1 Inhibitors and Lenvatinib for Intermediate and Advanced Hepatocellular Carcinoma After the Failure of Systemic Therapy Recommended by BCLC
Brief Title: HAIC in Combination with PD-1 Inhibitors and Lenvatinib for Intermediate and Advanced HCC After the Failure of Systemic Therapy Recommended by BCLC
Status: Recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Haibo Shao, Professor, MD, PhD, First Hospital of China Medical University
Other Study IDs: CHANCE2417
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: BCLC Stage B Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma; Hepatic Arterial Infusion Chemotherapy; Lenvatinib; PD-1; Systemic Therapy
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- HAIC plus Lenvatinib and PD-1 inhibitors: Each patient should receive at least 2 cycles of HAIC and 1cycles of PD-1 plus Lenvatinib. The interval between HAIC and Lenvatinib plus PD-1 inhibitors should be within 2 weeks.
  Interventions: Procedure: hepatic artery infusion chemotherapy; Drug: Lenvatinib + PD-1 monoclonal antibody

INTERVENTIONS:
Procedure: hepatic artery infusion chemotherapy — Hepatic arterial infusion chemotherapy including FOLFOX and RALOX
Drug: Lenvatinib + PD-1 monoclonal antibody — PD-1 inhibitors including Camrelizumab, Sintilimab, Tislelizumab

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of hepatic arterial infusion chemotherapy (HAIC) in combination with PD-1 inhibitors and Lenvatinib in patients with intermediate or advanced-stage hepatocellular carcinoma (HCC) after failure of systemic therapy recommended by BCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
2. Barcelona Clinic Liver Cancer (BCLC) stage C with the presence of portal vein tumor thrombus;
3. Has received previous systemic therapy recommended for HCC by BCLC, and the systemic therapy failed;
4. Both PD-1inhibitors and Lenvatinib patients received only include marketed drugs but are not limited to HCC approval;
5. HAIC was performed after the first PD-1 inhibitor/ Lenvatinib treatment or before treatment;
6. Received at least 2 cycles of HAIC；
7. Has repeated measurable intrahepatic lesions;
8. Child-Pugh class A or B.

Exclusion Criteria:

1. The interval between the failure of systemic therapy and the beginning of combination therapy longer than 3 months;
2. With other malignant tumors;
3. Unable to meet criteria of combination timeframe described above.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate or advanced HCC who have failed in systemic therapy recommended by BCLC and received HAIC in combination with PD-1 inhibitors and Lenvatinib under real-world practice conditions.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to approximately 2 years
  The OS is defined as the time from the initiation of any combination treatment to death due to any cause.

SECONDARY OUTCOMES:
Progression free survival(PFS) (Overall) | Up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease (according to mRECIST) or death due to any cause, whichever occurs first.
Progression free survival(PFS) of intra-hepatic lesions | Up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease of intra-hepatic lesions or death due to any cause, whichever occurs first.
Progression free survival(PFS) of extra-hepatic lesions | Up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented appearance of extra-hepatic lesions or death due to any cause, whichever occurs first.
Progression free survival(PFS) of portal vein tumor thrombus (PVTT) | Up to approximately 2 years
  The PFS is defined as the time from the initiation of any combination treatment to the first documented progressive disease of PVTT or death due to any cause, whichever occurs first.
Objective response rate(ORR) per RESCIST 1.1 | Up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per RECIST 1.1.
ORR per mRECIST | Up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented CR or PR per mRECIST.
ORR of PVTT | Up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented CR or PR of PVTT.
Adverse event(AE) per Common Terminology Criteria for Adverse Events(CTCAE) 5.0 | Up to approximately 2 years
  The percentage and degree of patients who experience at least one AE, whether or not considered related to the treatment, according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of China medical university, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided